CLINICAL TRIAL: NCT03899493
Title: Multichannel Surface Electromyography in Labor and Parturition
Brief Title: Electromyography in Labor and Parturition
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Kendra Gray, DO, Maternal Fetal Medicine Fellow, University of Arizona
Other Study IDs: 1809958902
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Labor
Keywords: Electroencephalography; Electromyography; Pelvic Floor; Labor curve; Intrauterine infection; Hypertensive Disorders of Pregnancy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primiparous & Multiparous: Women having borne at least one child > 20 weeks gestational age
  Interventions: Other: Observation
- Nulliparous: Women in whom this is their first pregnancy > 20 weeks who are anticipated to deliver
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Patients will be dispositioned to usual obstetric care which may include minimal intervention if spontaneous labor, induction of labor or augmentation of labor as indicated and dictated by the participants obstetrical provider. This study is observational only.

SUMMARY:
This study will examine how the uterus, abdominal wall, pelvic floor and brain interact during labor and parturition. It will uses electromyography (EMG) to compare the characteristics of the uterus, abdominal wall and perineum in subjects with and without various pregnancy characteristics.

EMG will help established burst frequency and characteristics of the uterus compared to other parts of the body during labor and delivery. Other parts of the body may include abdominal surfaces (for uterine, abdominal, maternal EMG and fetal heart rate monitoring), perineal surface (for perineal muscles monitoring) and the maternal scalp (brain monitoring). EEG measures the electrical activity of the brain. The activity is recorded using wire electrodes attached to the scalp or mounted on a cap placed on the head. E MG measures electrical activity from muscles. It uses wire electrodes placed on the skin over the muscles.

Pregnant adult volunteers and patients who present to the investigator's institution may be eligible for this study.

Participants will lay or sit in a semi-reclining chair with sticker electrodes placed on the body surface area of interest. Muscle and/or brain activity will be measured with EEG and EMG recordings.

DETAILED DESCRIPTION:
Objectives

* To define the relationship between uterine electrical activity EMG during labor and parturition to various phases of labor and cervical dilations.
* To define the relationship between uterine and body site electrical activity EMG and brain EEG during labor and parturition in patient with hypertensive disorders of pregnancy
* To characterize electrical activity of pelvic floor muscles in relationship to uterine and abdominal muscles during delivery between subsets of patients
* To examine the electrical activity of women in preterm labor and those with labor dystocias to observe the effects of various treatments, which may have an impact on preventing or augmenting labor progress.
* To observe the impact of naturally occurring pregnancy pathology and common obstetrical interventions on the changes in uterine, abdominal, pelvic floor and brain EEG/EMG characteristics as compared to health normal gravid patients.

Study Population:

Pregnant volunteers greater than 18 years of age who speak English.

Design:

During the course of the participant's admission, they will be dispositioned to usual obstetric care which may include minimal intervention if spontaneous labor, induction of labor or augmentation of labor as indicated. As part of the study protocol, enrolled participants will be monitored with external sensors/transducers. The device will be attached to a patient's body, which may include the abdominal surface, perineal surface and the mother's scalp by trained study staff through electrical leads that are connected to commercially available EMG or EEG electrodes that have adhesive material in contact with the surface of the patient. Recordings will be made at specific times during labor

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to the Labor & Delivery unit at Banner University Medical Center - Phoenix for either (a) labor or (b) induction of labor.
* Age > 18 years-old
* No contraindications to vaginal delivery

Exclusion Criteria:

* Non-English-speaking patients
* Known uterine abnormalities that may affect the normal contractility of the uterus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients eligible for inclusion in this study protocol will be aged 18 years-old and older, female, and pregnant. There will be no restrictions based on race or ethnic group beyond exclusion of non-English-speaking patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

PRIMARY OUTCOMES:
Burst Characteristic RMS | Through study completion, an average of 3 years
  EEG and EMG burst characteristics will be measured as RMS value (mV).
Burst Characteristic Median Frequency | Through study completion, an average of 3 years
  EEG and EMG burst characteristics will be measured as median frequency (Hz).
Burst Characteristic Duration | Through study completion, an average of 3 years
  EEG and EMG burst characteristics will be measured as duration (seconds).
Burst Characteristics Amplitude | Through study completion, an average of 3 years
  EEG and EMG burst characteristics will be measured as amplitude (mV).

CONTACTS AND LOCATIONS:
Overall Officials: Mike Foley, MD, Study Chair — BUMCP, Chair Department of Obstetrics and Gynecology; Kendra Gray, DO, Principal Investigator — Banner University Medical Center, MFM Fellow
Locations (1):
- Banner University Medical Center Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Creasy R, Resnik R, Iams J, Lockwood C, Moore T, Greene M. Creasy and Resnik's Maternal-Fetal Medicine, 7th Edition.; 2014. doi:10.1016/B978-1-4557-1137-6.00062-3
- [Result] Qian X, Li P, Shi SQ, Garfield RE, Liu H. Simultaneous Recording and Analysis of Uterine and Abdominal Muscle Electromyographic Activity in Nulliparous Women During Labor. Reprod Sci. 2017 Mar;24(3):471-477. doi: 10.1177/1933719116658704. Epub 2016 Jul 19. PMID 27436367
- [Result] Lucovnik M, Kuon RJ, Garfield RE. Assessment of parturition with cervical light-induced fluorescence and uterine electromyography. Comput Math Methods Med. 2013;2013:165913. doi: 10.1155/2013/165913. Epub 2013 Sep 29. PMID 24187578
- [Result] Trojner Bregar A, Lucovnik M, Verdenik I, Jager F, Gersak K, Garfield RE. Uterine electromyography during active phase compared with latent phase of labor at term. Acta Obstet Gynecol Scand. 2016 Feb;95(2):197-202. doi: 10.1111/aogs.12818. Epub 2015 Dec 8. PMID 26575523
- [Result] Lucovnik M, Trojner Bregar A, Bombac L, Gersak K, Garfield RE. Effects of vaginal progesterone for maintenance tocolysis on uterine electrical activity. J Obstet Gynaecol Res. 2018 Mar;44(3):408-416. doi: 10.1111/jog.13545. Epub 2018 Jan 3. PMID 29297950